CLINICAL TRIAL: NCT01855243
Title: Premix 70/30 Insulin Plus Supplemental Lunch Insulin in Comparison to Basal Plus Prandial Supplemental Scale and Sliding Scale Insulin in Hospitalized Patients With Type 2 Diabetes
Brief Title: Comparison on Efficacy and Safety of Three Inpatient Insulin Therapy in Type2 DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Said, Teaching Assistant, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CairoU teaching hospital
Record Dates: First submitted 2013-05-07; First posted 2013-05-16 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus (DM)
Keywords: Type 2 D M; sliding scale insulin; 70/30 insulin; basals insulin; supplemental insulin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin; Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- glargine plus supplemental glulisine (Active Comparator): Patients who will be recruited to be treated with glargine/glulisine, will received 50% of TDD as detailed demonstrated in Umpierrez et al., studies . as This includes administration of glargine (Lantus®) once every night plus glulisine (Apidra®) before each meal for BG ≥ 150 mg/dL. Glargine dose will be calculated as 0.2 U/kg/day for admission BG less than 200 mg/dL or 0.3 U/kg/day for BG exceeding 200 mg/dL. Glargine was given using Solostar Flex-Pen® once daily in the evening around 8:00 pm. Glulisine was given using the Solostar Flex-Pen® three times just before the meals for BG > 150 mg/dL according to hospital sliding scale. To avoid hypoglycemia, if for any reason, a subject missed a meal, the dose of glulisine will be held.
  Interventions: Drug: Glargine; Drug: glulisine
- 70/30 insulin plus supplemental lunch insulin (Active Comparator): Modified split-mixed insulin protocol adopted by Umpierrez et al., will be applied to patients treated with 70/30 insulin. Insulin dose will be started at 0.4 U/kg/day for admission BG less than 200 mg/dL or 0.5 U/kg/day for BG above 200 mg/dL. Two thirds of total daily dose (TDD)will be given before breakfast and 1/3 of TDD before dinner. Supplemental lunchtime regular insulin dose will given for BG > 150 mg/dL . Patients previously treated with 70/30 insulin before admission initially will receivethe same regimen as at in home.
  Interventions: Drug: regular insulin; Drug: 70/30 insulin
- Sliding Scale insulin (SSI) (Active Comparator): For SSI group, regular insulin will be administered three times daily subcutaneously approximately 30 min before meal for BG > 150 mg/dL (or every 8 hours if a patient was not eating) according to hospital sliding scale table
  Interventions: Drug: regular insulin

INTERVENTIONS:
Drug: regular insulin
  Arms: 70/30 insulin plus supplemental lunch insulin; Sliding Scale insulin (SSI)
Drug: 70/30 insulin
  Arms: 70/30 insulin plus supplemental lunch insulin
Drug: Glargine
  Other Names: lantus
  Arms: glargine plus supplemental glulisine
Drug: glulisine
  Other Names: apidra
  Arms: glargine plus supplemental glulisine

SUMMARY:
Purpose: To compare efficacy and safety of traditional sliding scale insulin (SSI) versus modified 70/30 insulin versus modified basal plus supplemental scale /bolus insulin regimens for glycemic control in hospitalized diabetic patients with diabetes.

Methods: In a prospective trial, patients with diabetes will be randomized to receive either traditional hospital SSI , or twice daily 70/30 insulin plus supplemental lunchtime insulin for BG ≥ 150 mg/dL or once every night glargine plus three times prandial glulisine for BG ≥ 150 mg/dL . 70/30 insulin and glargine will be started respectively at 0.4 and 0.2 U/kg/day for BG ≤ 200 mg/dL or 0.5 and 0.3 U/kg/day for BG above 200 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* known history of type 2 DM for longer than 3 months
* age between 18-64 year old,
* treatment with diet alone, any combination of oral antidiabetic agents and/or insulin before admission.

Exclusion Criteria:

* subjects with hyperglycemia without any known history of DM
* presence of diabetic ketoacidosis (DKA)
* patients admitted to intensive care unit (ICU)
* subjects expected to undergo surgery during the hospitalization course
* patients with clinically relevant hepatic disease impaired renal function (serum creatinine ≥ 3.0 mg/dL) systemic infections pregnancy patients on medications known to interfere with the blood glucose level (either increasing or decreasing

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- the department of internal medicine, Cairo University teaching hospitals,, Cairo, Egypt

REFERENCES:
- [Background] Umpierrez GE, Smiley D, Zisman A, Prieto LM, Palacio A, Ceron M, Puig A, Mejia R. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes (RABBIT 2 trial). Diabetes Care. 2007 Sep;30(9):2181-6. doi: 10.2337/dc07-0295. Epub 2007 May 18. PMID 17513708
- [Background] Umpierrez GE, Hor T, Smiley D, Temponi A, Umpierrez D, Ceron M, Munoz C, Newton C, Peng L, Baldwin D. Comparison of inpatient insulin regimens with detemir plus aspart versus neutral protamine hagedorn plus regular in medical patients with type 2 diabetes. J Clin Endocrinol Metab. 2009 Feb;94(2):564-9. doi: 10.1210/jc.2008-1441. Epub 2008 Nov 18. PMID 19017758

RESULTS

PARTICIPANT FLOW:
Recruitment Details: a known history of type 2 DM for longer than 3 months admitted to general medicine wards, age between 18 - 64 year old, treatment with diet alone, any combination of oral antidiabetic agents and/or insulin before admission.
Groups:
- Glargine Plus Supplemental Glulisine: Patients who will be recruited to be treated with glargine/glulisine, will received 50% of TDD as detailed demonstrated in Umpierrez et al., studies . as This includes administration of glargine (Lantus®) once every night plus glulisine (Apidra®) before each meal for BG ≥ 150 mg/dL. Glargine dose will be calculated as 0.2 U/kg/day for admission BG less than 200 mg/dL or 0.3 U/kg/day for BG exceeding 200 mg/dL. Glargine was given using Solostar Flex-Pen® once daily in the evening around 8:00 pm. Glulisine was given using the Solostar Flex-Pen® three times just before the meals for BG > 150 mg/dL according to hospital sliding scale. To avoid hypoglycemia, if for any reason, a subject missed a meal, the dose of glulisine will be held.
  Glargine
  glulisine
- 70/30 Insulin Plus Supplemental Lunch Insulin: Modified split-mixed insulin protocol adopted by Umpierrez et al., will be applied to patients treated with 70/30 insulin. Insulin dose will be started at 0.4 U/kg/day for admission BG less than 200 mg/dL or 0.5 U/kg/day for BG above 200 mg/dL. Two thirds of total daily dose (TDD)will be given before breakfast and 1/3 of TDD before dinner. Supplemental lunchtime regular insulin dose will given for BG > 150 mg/dL . Patients previously treated with 70/30 insulin before admission initially will receivethe same regimen as at in home.
  regular insulin
  70/30 insulin
- Sliding Scale Insulin (SSI): For SSI group, regular insulin will be administered three times daily subcutaneously approximately 30 min before meal for BG > 150 mg/dL (or every 8 hours if a patient was not eating) according to hospital sliding scale table
  regular insulin
Period: Overall Study
Arm/Group | Glargine Plus Supplemental Glulisine | 70/30 Insulin Plus Supplemental Lunch Insulin | Sliding Scale Insulin (SSI)
Started | 20 | 21 | 22
Completed | 19 | 21 | 22
Not Completed | 1 | 0 | 0
Not completed — develpoed diabetic ketoacidosis | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glargine Plus Supplemental Glulisine | 70/30 Insulin Plus Supplemental Lunch Insulin | Sliding Scale Insulin (SSI) | Total
Number analyzed (Participants) | 19 | 21 | 22 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11) | 55 (7) | 55 (7) | 55 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 15 | 41
  Male | 5 | 9 | 7 | 21
Region of Enrollment [Number; unit: participants]
  Egypt | 19 | 21 | 22 | 62
Body weight [Mean (Standard Deviation); unit: Kg] | 75 (11) | 78 (20) | 73 (12) | 76 (15)
BMI [Mean (Standard Deviation); unit: Kg/m2] | 31 (6) | 31 (7) | 31 (5) | 31 (5)

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Blood Glucose (BG) Concentration During Their Hospital Stay.
Time Frame: during hospital stay which is expected to be average 3 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Glargine Plus Supplemental Glulisine | 70/30 Insulin Plus Supplemental Lunch Insulin | Sliding Scale Insulin (SSI)
Number analyzed (Participants) | 19 | 21 | 22
mg/dL | 221 (67) | 179 (36) | 222 (67)

2. Secondary Outcome: Number of Patients Developed Hypoglycemic Events
Description: Hypoglycemic episodes are classified as major (BG ≤ 40 mg/dL or associated with impaired mental status or loss of consciousness), or minor (BG between 40 and 59 mg/dL) events.
Time Frame: during hospital stay which is expected to be average 3 weeks
Measure: Number; unit: participants
Arm/Group | Glargine Plus Supplemental Glulisine | 70/30 Insulin Plus Supplemental Lunch Insulin | Sliding Scale Insulin (SSI)
Number analyzed (Participants) | 19 | 21 | 22
participants
  Minor (BG between 40 - 59 mg/dL | 3 | 0 | 1
  Major (BG ≤ 40 mg/dL) | 2 | 0 | 0

3. Secondary Outcome: Number of Patients Developed Episodes of Severe Hyperglycemia
Description: Hyperglycemic events are defined as BG > 300 mg/dL.
Time Frame: during hospital stay which is expected to be average 3 weeks
Measure: Number; unit: participants
Arm/Group | Glargine Plus Supplemental Glulisine | 70/30 Insulin Plus Supplemental Lunch Insulin | Sliding Scale Insulin (SSI)
Number analyzed (Participants) | 19 | 21 | 22
participants | 10 | 4 | 15

4. Secondary Outcome: Mortality Rate
Time Frame: during the hospital stay which is expected to be average 3 weeks
Measure: Number; unit: participants
Arm/Group | Glargine Plus Supplemental Glulisine | 70/30 Insulin Plus Supplemental Lunch Insulin | Sliding Scale Insulin (SSI)
Number analyzed (Participants) | 19 | 21 | 22
participants | 0 | 0 | 0

5. Primary Outcome: Mean BG After First Day of Hospitalization
Time Frame: after first day of hospitalization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Glargine Plus Supplemental Glulisine | 70/30 Insulin Plus Supplemental Lunch Insulin | Sliding Scale Insulin (SSI)
Number analyzed (Participants) | 19 | 21 | 22
mg/dL | 225 (65) | 171 (38) | 218 (71)

ADVERSE EVENTS:
Time Frame: during hospital stay which is expected to be 3 weeks
Description: Major hypoglycemia (BG ≤ 40 mg/dL) associated with impaired mental status or loss of consciousness
Arm/Group | Glargine Plus Supplemental Glulisine | 70/30 Insulin Plus Supplemental Lunch Insulin | Sliding Scale Insulin (SSI)
Serious Adverse Events (participants affected / at risk) | 2/19 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 10/19 | 4/21 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine Plus Supplemental Glulisine (N=19) | 70/30 Insulin Plus Supplemental Lunch Insulin (N=21) | Sliding Scale Insulin (SSI) (N=22)
major hypoglycemia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) — Major Hypoglycemic episodes (BG ≤ 40 mg/dL or associated with impaired mental status or loss of consciousness
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine Plus Supplemental Glulisine (N=19) | 70/30 Insulin Plus Supplemental Lunch Insulin (N=21) | Sliding Scale Insulin (SSI) (N=21)
Severe Hyperglcemia eposide (Nervous system disorders) | 10 (22) | 4 (8) | 15 (30) — severe hyperglycemia episode (BG > 300 mg/dL)

LIMITATIONS AND CAVEATS:
self funded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No